CLINICAL TRIAL: NCT07233486
Title: A Multicenter, Randomized, Crossover Clinical Trial Study of Digital Intelligence Software in Patients With MAFLD
Acronym: DISMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025(E2)-HS-053; 2023ZD0508704 (Other Grant/Funding Number: Noncommunicable Chronic Diseases-National Science and Technology Major Project)
Record Dates: First submitted 2025-08-28; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: MAFLD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Life intervention group (No Intervention): Detailed nutritional intervention protocols were developed according to patients' food preferences, dietary habits, physical activity levels, working conditions, sociocultural conditions, and lifestyle. Low-carbon diet and balanced diet were adopted for dietary intervention. According to the patients' basic metabolic level, overweight and fatty liver degree, a calorie restriction diet was formulated, and it was recommended to reduce 500-1000 kcal calories per day, a balanced diet of pastries and carbohydrates, with increased intake of whole grains, omega-3 fatty acid, and dietary fiber. Choose the right ingredients for your particular patient's diet
- Digital Intelligence Software Group (Placebo Comparator): Study participants were guided by the program officer to download and register the"Data Intelligence software (patient-side)" and to establish a relationship with the clinicians involved in the study, baseline data were collected under the guidance of the program director, health records were created, and data were collected using a software-supported"Body composition analyzer.". The participating clinicians evaluated the subjects through the"Digital Intelligence software (doctor side)", and formulated the diet and exercise program according to the individual conditions of the subjects.
  Interventions: Procedure: Digital Intelligence Software Intervention Group

INTERVENTIONS:
Procedure: Digital Intelligence Software Intervention Group — Study participants were guided by the program officer to download and register the"Data Intelligence software (patient-side)" and to establish a relationship with the clinicians involved in the study, baseline data were collected under the guidance of the program director, health records were created, and data were collected using a software-supported"Body composition analyzer.". The participating clinicians evaluated the subjects through the"Digital Intelligence software (doctor side)", and formulated the diet and exercise program according to the individual conditions of the subjects.
  Arms: Digital Intelligence Software Group

SUMMARY:
Cirrhosis associated with metabolic associated fatty liver disease (MAFLD) can lead to a series of adverse outcomes in and outside the liver, but there is no approved treatment so far. In recent years, the prevalence of MAFLD-related cirrhosis in our country is increasing rapidly, but its clinical, pathological characteristics and natural prognosis are not clear, and there is a lack of standardized and effective prevention and treatment strategies.Through"Digital Intelligence software" to assist clinicians in MAFLD patients with remote data intervention, lifestyle intervention guidance and follow-up management, to evaluate the efficacy and safety of the intervention software on body weight and blood glucose in patients with MAFLD.

ELIGIBILITY:
Inclusion Criteria

1. Adult patients aged 18-65 years with a BMI of 24-35 kg/m².
2. Confirmed diagnosis of Metabolic-associated Fatty Liver Disease (MAFLD), defined by a FibroScan® result > 248 dB/m or an MRI-PDFF > 5%.
3. Willing and able to provide written informed consent and comply with the study protocol, including the use of a compatible smartphone for digital health components.
4. If treated for Type 2 Diabetes Mellitus (T2DM), must be on a stable medication regimen for at least 3 months prior to baseline (Day 0), with the expectation to maintain stability throughout the study barring medical necessity.
5. If taking medications with potential NASH-remitting effects (e.g., vitamin E, thiazolidinediones), must be on a stable dose for at least 3 months prior to Day 0.

Exclusion Criteria

1. Subjects were excluded from participation if they met any of the following criteria, based on the most recent pre-randomization assessments:
2. Evidence of cirrhosis, defined as histological stage F4 or its clinical equivalent.
3. History of heavy alcohol consumption (>30 g/day for males, >20 g/day for females) for more than 3 consecutive months within one year prior to screening.
4. Prior or planned solid organ transplantation (excluding corneal transplants).
5. Planned bariatric surgery. A history of bariatric surgery was permitted only if weight had been stable (variation <10%) for at least 3 months prior to screening.
6. Presence of other chronic liver diseases, including:
7. Hepatitis B surface antigen (HBsAg) positivity.
8. Hepatitis C virus (HCV) RNA positivity.
9. Primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis, or overlap syndromes.
10. Wilson's disease, alpha-1 antitrypsin deficiency (ZZ phenotype), or hereditary hemochromatosis.
11. History of Type 1 Diabetes Mellitus. Uncontrolled Type 2 Diabetes Mellitus, defined as HbA1c >9% or current insulin therapy.
12. History of hepatic decompensation events (e.g., ascites, hepatic encephalopathy, variceal hemorrhage).
13. Any of the following laboratory abnormalities at screening:
14. Platelet count < 150,000/mm³
15. Albumin < 3.0 g/dL
16. International Normalized Ratio (INR) > 1.3
17. Alkaline Phosphatase (ALP) > 2 × Upper Limit of Normal (ULN)
18. Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) > 5 × ULN
19. Total Bilirubin > 1.3 × ULN (except in cases of documented Gilbert's syndrome)
20. Estimated Glomerular Filtration Rate (eGFR) < 60 mL/min/1.73 m²
21. Hemoglobin < 10 g/dL
22. Uncontrolled thyroid dysfunction, defined as a thyroid-stimulating hormone (TSH) level < 0.1 or > 10 µIU/mL at screening.
23. Documented HIV-1 or HIV-2 infection.
24. Known Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency.
25. Significant cardiovascular history, including myocardial infarction, unstable angina, heart failure, uncontrolled arrhythmia, coronary artery bypass graft, or percutaneous coronary intervention within one year prior to screening.
26. Diagnosis of malignancy within the past 2 years (except for adequately treated basal cell carcinoma or cutaneous squamous cell carcinoma).
27. Severe co-morbid respiratory, cardiac, cerebrovascular, hepatic, or renal conditions that, in the investigator's judgment, would preclude safe participation in a diet and exercise intervention.
28. Active, severe infection requiring parenteral antimicrobial therapy within 30 days of screening.
29. Major surgery within 30 days prior to screening.
30. Chronic use of medications known to promote hepatic steatosis (e.g., systemic corticosteroids, amiodarone, methotrexate, tamoxifen, valproic acid) within 3 months of screening. Short-term, low-dose corticosteroid use was permissible.
31. Current or planned treatment with radiation therapy, cytotoxic chemotherapy, or immunomodulatory agents (e.g., interleukins, interferons).
32. Treatment with any investigational agent within 6 months prior to screening, or prior participation in a clinical trial for NASH/MAFLD within 6 months.

Pregnancy or lactation.

1.Any other condition or circumstance that, in the opinion of the Investigator, would compromise patient safety or the validity of the study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Body weight | 48weeks
  Absolute and relative changes from baseline in body weight

SECONDARY OUTCOMES:
Fasting plasma glucose | 48week
  Compare the changes in fasting blood glucose before and after treatment
Liver MRI PDFF | 48weeks
  To evaluate the effects of weight and glucose reduction interventions on proton density fat fraction (MRI-PDFF) in patients with MAFLD
Liver FibroScan | 48week
  liver fat attenuation parameter (CAP) , liver stiffness value (LSM)
Body Mass Index (BMI) | 48week
  Clarify how multiple measurements will be aggregated to arrive at one reported value weight and height will be combined to report BMI in kg/m^2)

OTHER OUTCOMES:
Biochemical indicators | 48week
  Serum levels of aspartate aminotransferase (AST U/L) and alanine aminotransferase (ALT U/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Normal University Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The study has not been completed